CLINICAL TRIAL: NCT04103164
Title: Open Label, Prospective, Single-Center Pilot Study to Evaluate the Effect of Multiple Passes on Port Wine Stain Treatments With the Cutera Excel V™ Laser.
Brief Title: Pilot Study to Evaluate the Effect of Multiple Passes on Port Wine Stain Treatments With the Cutera Excel V™ Laser.
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: The laser is currently being worked on
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Richard Rox Anderson, MD, Director of Wellman Center for Photomedicine, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018P000366
Record Dates: First submitted 2018-05-23; First posted 2019-09-25 (Actual); Last update posted 2019-10-15 (Actual); Status verified 2019-10

CONDITIONS: Port-Wine Stain
MeSH Terms: conditions — Port-Wine Stain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Cutera® excel V laser arm (Experimental): After the PWS is be divided into five equal portions, four of those portions treated once with a different laser fluence using the multiple-pass approach (2 J/cm² vs 4 J/cm² vs 6 J/cm² vs 8 J/cm²), and one of the portions treated with single-pass approach at 8 J/cm²
  Interventions: Device: Cutera excel V™ Laser

INTERVENTIONS:
Device: Cutera excel V™ Laser — The Cutera® excel V laser is manufactured by Cutera, Inc. This laser with 532 nm KTP and 1064 nm Nd:YAG wavelengths has received 510(k) clearance by the U.S. Food and Drug Administration (FDA) to market the device for use in surgical and aesthetic applications requiring selective photothermolysis of target chromophores in soft tissue 510(k) number 022226. The 532 nm wavelength is indicated for the coagulation and hemostasis of benign vascular and cutaneous lesions in dermatology including, but not limited to, benign vascular lesions like angiomas, hemangiomas, port wine stains, venous anomalies and telangiectasia; benign pigmented lesions like nevi, lentigines, chloasma, café-au-lait; verrucae; skin tags; keratoses; plaques. The Cutera® excel V laser has also obtained the European CE Mark. The system was tested to ensure compliance with federal laser performance standards as applicable.

SUMMARY:
Two limitations of single pulse, laser treatment of port-wine stains (PWS) are: (i) hemorrhage and purpura which may lead to post-treatment pigmentation and (ii) the necessity for repeated treatment sessions. In contrast, multiple pulses induce summation of irreversible, thermal injury from a series of lower-peak temperature heating cycles and may therefore reduce mechanical injury while preserving the selectivity of photothermal injury. Ideally, hemorrhage could be prevented and the efficiency of vessel closure could be greater. A clinical and histological pilot study of 10 adults with either facial or non-facial PWS is therefore proposed here.

ELIGIBILITY:
Inclusion Criteria:

Subject must be able to read, understand and sign the Informed Consent Form. Female or Male, 18 to 65 years of age (inclusive). Fitzpatrick Skin Type I - VI. Have either facial or non-facial port wine stain covering at least 50cm² area on the body.

Must be willing to have Cutera excel V laser treatments (532 nm) with prototype EV handpiece and PWS scanner and able to adhere to the treatments, follow-up visit schedule, and post-treatment care instructions.

Willing to have very limited sun exposure and use sunscreen on the treatment area every day for the duration of the study, including the follow-up period.

Willing to have digital photographs taken of the treatment area and agree to use of photographs for presentation (educational and/or marketing), publications, and any additional marketing purposes.

Agree to not undergo any other cosmetic procedure(s) or treatment(s) on the face during the study and has no intention of having such procedures performed during the course of the study.

For female subjects: not pregnant or lactating and is either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study.,

Exclusion Criteria:

Participation in a clinical trial of another drug, or device administered to the treatment area, within 3 months prior to enrollment or during the study.

Any type of prior cosmetic or port wine stain treatment to the target area within 3 months of study participation.

Suffering from significant skin conditions in the treated areas or inflammatory skin conditions, including but not limited to, open lacerations or abrasions, hidradenitis, rash, infection , or dermatitis of the treatment area prior to treatment (duration of resolution as per the Investigator's discretion).

Pregnant and/or breastfeeding, or planning to become pregnant. Significant concurrent illness, such as diabetes mellitus, immunosuppression/immune deficiency disorders (including HIV infection or AIDS) or using immunosuppressive medication.

Hypersensitivity to light exposure. Any use of medication that is known to increase sensitivity to light according to the Investigator's discretion.

History of keloid scarring, hypertrophic scarring or abnormal wound healing or prone to bruising.

Has a history of squamous cell carcinoma or melanoma in the treatment area. History of epidermal or dermal disorders (particularly if involving collagen or microvascularity), including collagen vascular disease or vasculitic disorders.

A history or active skin condition that in the opinion of the Investigator may interfere/confound with the treatment.

History of connective tissue disease, such as systemic lupus erythematosus or scleroderma.

History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen.

History of pigmentary disorders, particularly tendency for hyper- or hypo-pigmentation, or any that are considered not acceptable by the study investigator.

Excessively tanned or active sun tan in facial area to be treated, or unable/unlikely to refrain from tanning during the study.

Excessive facial hair in the area to be treated (beards, sideburns, and/or moustache,) that would interfere with diagnosis, assessment, and treatment.

As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study, including excessive alcohol or drug abuses, or a condition that would compromise the subject's ability to comply with the study requirements.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2020-01-15 (Estimated); Primary Completion 2020-07-15 (Estimated); Study Completion 2020-07-15 (Estimated)

PRIMARY OUTCOMES:
Optimal Fluence based on efficacy and safety measurements using photographs | 6 months
  Find the optimal fluence in a multiple split port wine stain treatment, with 2 J/cm2 (low fluence control) vs 4 J/cm2 vs 6 J/cm2 vs 8 J/cm2 in the multiple-pass approach, compare it to our standard single-pass approach at 8 J/cm2.
  -The efficacy of treatment assessed by improvement in PWS among the 5 treated areas using before and after digital photographic assessment. Each digital photographic image will include a color card, so that changes can be compared from day 0 to final visit.
  The hypothesis is that the effect of multiple passes on Port Wine Stain treatments with the Cutera excel V™ Laser would be more effective than the current single pass treatment.

SECONDARY OUTCOMES:
Optimal Fluence based on efficacy and safety measurements using questionnaires/surveys. | 6 months
  - Safety will be assessed by questionnaires/surveys about frequency and severity of post treatment side-effects among the 5 treated areas after one treatment throughout the study, such as using the Visual Analog Score for Pain.
  The hypothesis is that the effect of multiple passes on Port Wine Stain treatments with the Cutera excel V™ Laser would be more safe than the current single pass treatment.

OTHER OUTCOMES:
Histologic differences in microvasculature post-treatment based on punch biopsies | 6 months
  • Compare histology among the 5 treated areas after treatment to evaluate the differences in microvasculature.
  - This will be done by obtaining punch biopsies from the different treated areas and analyzing the histological slides for differences in microvasculature.

CONTACTS AND LOCATIONS:
Overall Officials: Rox Anderson, MD, Principal Investigator — MGH
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Reddy KK, Brauer JA, Idriss MH, Anolik R, Bernstein L, Brightman L, Hale E, Karen J, Weiss E, Elston D, Geronemus RG. Treatment of port-wine stains with a short pulse width 532-nm Nd:YAG laser. J Drugs Dermatol. 2013 Jan;12(1):66-71. PMID 23377330
- [Background] Jacobs AH, Walton RG. The incidence of birthmarks in the neonate. Pediatrics. 1976 Aug;58(2):218-22. PMID 951136